CLINICAL TRIAL: NCT03998358
Title: Characterization of Fatigue in Military Personnel With Traumatic Brain Injuries
Status: Withdrawn | Type: Observational
Why Stopped: Recruitment method is no longer active.
Sponsor: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 190115; 19-NR-0115
Record Dates: First submitted 2019-06-25; First posted 2019-06-26 (Actual); Last update posted 2021-03-25 (Actual); Status verified 2021-03

CONDITIONS: Traumatic Brain Injury; Neurobehavioral Manifestation; Sleep Disorder; Fatigue
Keywords: Circadian Rhythm; Biomarkers; Neuroendocrine; Sleep; Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic; Neurobehavioral Manifestations; Sleep Wake Disorders; Fatigue

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood and PBMCs

GROUPS / COHORTS (2):
- High Fatigue: TBI patients with significant fatigue as calculated by a score of >= 5.5 on the Fatigue Severity Scale
- Low Fatigue: TBI patients without significant fatigue as calculated by a score of < 5.5 on the Fatigue Severity Scale

SUMMARY:
Background:

People who have had a traumatic brain injury (TBI) often experience fatigue. Fatigue is the feeling tired all the time. Researchers want to learn more about how TBI and fatigue are related.

Objective:

To better understand fatigue after TBI in active duty military and veterans.

Eligibility:

Active duty service members or veterans ages 25-40 who have sustained at least 1 TBI more than 6 months but less than 5 years ago

Design:

Participants will be screened with:

* Medical history
* Physical exam
* Blood and urine tests

Participants will have Visit 1 the same day as screening. This will include questionnaires and interviews. These will be about their fatigue, quality of life, and health.

Participants will wear an activity monitor on their wrist and complete a sleep diary for 7 days at home.

Participants will have Visit 2: They will stay in the clinic for 2 nights. The visit will include:

* Tests of memory, attention, and thinking
* Placement of intravenous (IV) line: A needle will guide a thin plastic tube into the participant s arm vein.
* 2 overnight sleeps tests: Participants brain waves will be recorded while they sleep. Small electrodes will be placed on the scalp. Monitors will be placed on the skin. These will measure breathing, heart rate, and movement. Blood will be drawn overnight through the IV line.
* Optional hydrocortisone stimulation test: Participants will receive the hormone through the IV line. Blood will be drawn through the IV line 5 times over 1 hour.
* Optional MRI: Participants will lie in a machine. This machine is a metal cylinder that takes pictures of the brain.

DETAILED DESCRIPTION:
Objective: Traumatic brain injury (TBI) is the signature injury of recent wars. Fatigue is a pervasive and debilitating consequence of TBIs, experienced by up to 80% of military personnel following TBI. If present greater than 6 months post-injury, fatigue is classified as chronic and may hinder recovery and affect return to service in military personnel. However, the pathophysiology through which TBI results in fatigue symptomology remains unclear. This protocol will examine several pathways that have been hypothesized to underlie the association between TBI and fatigue including; sleep disturbances, neuroendocrine and mitochondrial abnormalities. Sleep disturbances and fatigue overlap and frequently co-occur after TBI. However, to date no published studies have investigated the association between objectively measured sleep and fatigue following TBI with and without significant fatigue in military personnel. The second pathway involves dysfunction of the neuroendocrine system, which participates in the regulation of sleep states, circadian function, and attention. Deficits in neuroendocrine function, including putative changes in crucial neuronal populations in the hypothalamus and in somatotrophic cells of the anterior pituitary will result in changes in regulatory hormones such as growth hormone (GH). Evidence suggests that disruptions to GH may be associated with fatigue, however, current findings are mixed. The final pathway may be through mitochondrial dysfunction. Early results from multiple fields have shown that decreased mitochondrial markers have been associated with fatigue, however few studies have looked at these predicted associations in TBI populations. It is evident that further research is needed to examine the relationships between TBI and fatigue. Thus, this protocol aims to identify the pathways associated with TBI and fatigue. Findings from this protocol may lead to novel targets for intervention and reduction of fatigue symptomology following TBI.

Aim: To identify factors that are associated with the persistence of fatigue symptomology, at or greater than 6 months post TBI.

Protocol population: Up to 74 military personnel will be recruited into this protocol. All participants will have experienced their most recent TBI >= 6 months and <= 5 years prior to protocol participation.

Design: We will compare military personnel who have sustained a TBI with and without subsequent fatigue symptomology. This protocol will have two visits, one outpatient and one inpatient to NIH which include:

Screening Visit: All participants will undergo a clinical evaluation of TBI history, fatigue, and complete self-report questionnaires. Participants will also be given an actigraph and sleep diary to take home and complete.

Sleep Visit: All participants will undergo two, consecutive, overnight polysomnography (PSG) tests, which includes one night of serial blood sampling to examine endocrine function and neuropeptide release. Over the two days, participants may also complete an optional hydrocortisone stimulation test and their mitochondrial respiratory profile will be assessed. During this in-patient stay, all participants will undergo neurocognitive testing and have an opportunity to undergo magnetic resonance imaging (MRI).

ELIGIBILITY:
* INCLUSION CRITERIA:
* Are 25 to 40 years of age
* Are active duty service members or veterans
* May be NIH employees/staff who are either active duty service members or veterans; except for those who are employed by NINR or subordinates, relatives, and/or co-workers of NINR employees/staff
* Have sustained at least 1 TBI, >= 6 months and <= 5 years since their most recent TBI, which includes any self-reported loss of consciousness (LOC) established by the OSU during the pre-screening phone call
* Are able to provide their own consent
* Are able to understand the protocol, as shown by scoring a 6 out of 6 on a consent quiz

EXCLUSION CRITERIA:

* Currently receiving treatment for a medical illness or recent injury that precludes protocol participation, may interfere with study participation, and/or should be treated/stabilized prior to study participation for safety reasons (e.g., cancer, recent fracture(s) requiring therapy and/or pain medication, severe infection). Individuals with stable medical conditions such as hypertension that are controlled by medication will be included.
* Current physical health status will be assessed by self-report, history and physical exam by a credentialed physician or nurse practitioner, and standard laboratory tests.
* Current unstable endocrine disorder (e.g., uncontrolled diabetes). Unstable endocrine disorders require treatment to ensure health and safety of the patient before participation is possible. Individuals with stable endocrine disorders (e.g., controlled diabetes) may participate in the protocol but they will be excluded from the hydrocortisone stimulation test. This will be assessed by self-report during the history and physical exam and by standard laboratory tests.
* Have a major medical illness that is associated with fatigue (e.g., chronic fatigue [diagnosed prior to their TBI or less than 6 months following TBI], multiple sclerosis, or cancer). This will ensure that symptoms of fatigue are as a result of TBI and not another co-morbid illness. This will be assessed by self-report.
* Currently consuming any of the following sleep modifying medications: benzodiazepines; benzodiazepine receptor agonists; opiates; or sedatives. These medications will directly affect the results of the PSG and actigraphy analysis, as such participants currently taking these medications will be excluded. This will be assessed by self-report.
* Currently using the sleep modifying medications melatonin and/or Benadryl greater than 2 times per week and/or unable or unwilling refrain from using them during protocol participation. These medications will directly affect the results of the PSG and actigraphy analysis, as such participants who are unwilling/unable to refrain from using these medications will be excluded. This will be assessed by self-report.
* Current psychiatric condition for which immediate treatment is required to prevent harm to self or others such as active suicidality or active manic phase in someone who has bi-polar disorder. This is to ensure patient safety and care. This will be assessed by self-report and as part of the history and physical exam.
* Are pregnant. Pregnancy is associated with increased fatigue and sleep disturbances, as such this condition will affect the outcomes of this analysis.his will be assessed by self-report. This will also be assessed on visit 2 by a urine pregnancy test. Individuals who are nursing are eligible but will not participate in the hydrocortisone stimulation test.
* Received a diagnosis of severe obstructive sleep apnea (OSA) and/or current reliance on continuous positive airway pressure (CPAP) therapy to aid sleep. Severe OSA and CPAP use will directly affect the result s of this study, as such these participants will be excluded. This will be assessed by self-report.

  **Participant may be able to participate in the protocol but will not be able to have an MRI if they have any of the following:
* Metal in the body such as pacemakers, stimulators, pumps, aneurysm clips, metallic prostheses, artificial heart valves, cochlear implants or shrapnel fragments, or if they are a welder or metal worker
* Claustrophobia
* Are not able to lie comfortably flat on their back for up to 60 minutes

  **Participant may be able to participate in the protocol but will not be able to have the hydrocortisone stimulation test if they have any of the following:
* History of endocrine disorder or dysfunction (including thyroid, adrenal, pancreatic and pituitary disorders)
* Abnormal lab values that may indicate endocrine disorder or dysfunction
* Mother who is currently nursing an infant

Ages: 25 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Up to 74 military personnel will be recruited into this protocol. All participants will have experienced their most recent TBI >= 6 months and <= 5 years prior to protocol participation.@@@@@@
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-03-19 (Actual); Primary Completion 2021-03-19 (Actual); Study Completion 2021-03-19 (Actual)

PRIMARY OUTCOMES:
Determine differences in objective sleep measures determined by actigraphy and PSG data in military personnel with and without fatigue following a TBI. | Study completion
  The PSG will be scored by the Clinical Center Sleep Service within two weeks and will generate the following data: -Sleep Onset Latency (SOL): Is a measurement of the time taken to fall asleep from the time the lights were turned off. On average, this process takes approximately 20 minutes. - Sleep efficiency (SE): the number of minutes of sleep divided by the number of minutes in bed. Normal is approximately 85 to 90% or higher, but in-lab values are often less. -Sleep stages; From this information each 30-second epoch is scored as "awake" or one of 4 sleep stages: 1, 2, 3, and REM or Rapid Eye Movement sleep. Stages 1-3 are together called non-REM sleep. Non-REM sleep is distinguished from REM sleep, which is altogether different. Delta power for each stage will also be examined. The primary outcome being assessed will be delta power of SWS and REM between fatigued and non-fatigued.

SECONDARY OUTCOMES:
Determine differences in neurobehavioral and neurocognitive functioning in military personnel with and without fatigue following a TBI. | Study Completion
  Determine differences in neurobehavioral and neurocognitive functioning in military personnel with and without fatigue following a TBI
Describe differences in plasma concentration levels of neuroendocrine proteins during overnight hours in military personnel with and without fatigue following a TBI. | Study Completion
  Describe differences in plasma concentration levels of neuroendocrine proteins during overnight hours in military personnel with and without fatigue following a TBI.
Determine differences in neuroendocrine and mitochondrial functionality in military personnel with and without fatigue following a TBI. | Study Completion
  Determine differences in neuroendocrine and mitochondrial functionality in military personnel with and without fatigue following a TBI.
Compare group differences in level of fatigue between the two protocol visits. | Study Completion
  Compare group differences in level of fatigue between the two protocol visits.
Determine differences in perceived sleep quality (PSQI) and actual sleep quality as measured by actigraphy. | Study Completion
  Determine differences in perceived sleep quality (PSQI) and actual sleep quality as measured by actigraphy.
Compare volume of hypothalamus, attentional + arousal regions of interest as well as fractional anisotropy (FA), axial diffusivity (AD), radial diffusivity and white matter integrity using DTI in military personnel w and w/out fatigue following ... | Study Completion
  Compare volume of hypothalamus, attentional + arousal regions of interest as well as fractional anisotropy (FA), axial diffusivity (AD), radial diffusivity and white matter integrity using DTI in military personnel w and w/out fatigue following a TBI.
Determine if there are group differences in actigraphically measured sleep, light, and physical activity. | Study Completion
  Determine if there are group differences in actigraphically measured sleep, light, and physical activity.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Gill, Ph.D., Principal Investigator — National Institute of Nursing Research (NINR)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2019-NR-0115.html